CLINICAL TRIAL: NCT03123679
Title: The Added Value of Quantification of Lung Function in Patients Undergoing Radiotherapy, Using Tc-99m-MAA SPECT-CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-17-ES-0723-CTIL
Record Dates: First submitted 2017-04-02; First posted 2017-04-21 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: pulmonary perfusion/reserve with Tc-99m-MAA SPECT/ Low dose CT — 1. Patient referred to radiotherapy treatment are evaluated with a baseline PFT [Forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC), diffusing capacity of the lung for carbon monoxide (DLCO), Alveolar gas volume (VA)].
  2. RT simulation at the radiotherapy department and treatment planning.
  3. Baseline evaluation of pulmonary perfusion/reserve with Tc-99m-MAA SPECT/ Low dose CT.
  4. Radiotherapy.

SUMMARY:
Adult patients referred to radiotherapy treatment of primary or secondary malignant involvement of the lung parenchyma, who are not meeting the exclusion criteria, will be introduced to the study and suggested to participate in it by the radiotherapist, Dr Viacheslav Soyfer, M.D. from the Institute of Radiotherapy Tel Aviv (Sourasky) Medical Center.

They will sign an informed consent and the study will be conducted based on the agreement of the institutional ethical committee, prior to perfusion study.

Each patient will be evaluated three times: prior to treatment, a baseline evaluation mid-follow-up period 6 weeks post initiation of radiotherapy and a delayed follow up 6 months post treatment. Each SPECT/ Low dose CT assessment will take place within two weeks of the clinical and PFT assessment.

The study will take place within a duration of two years, from recruiting the participating patients to the completion of the study protocol by the last recruited patient. For the individual patient, the duration of participation is six months.

Perfusion SPECT/ Low dose CT studies with a non-diagnostic low dose chest CT will be performed after the I.V. injection of 4 mCi 99m-Tc-MAA. SPECT/ Low dose CT scan will be acquired immediately post injection on a GE OPTIMA NM/CT 640 camera. In order to obtain a better definition of the irradiated fields, we will co-register the SPECT/ Low dose CT with high-resolution CT provided from the Institute of Radiotherapy. In this procedure, the low dose chest CT is used as a bridge between high resolution CT and the functional imaging SPECT. Using the Q.Lung segmentation tool, individual whole lung function and lung subunits will be assessed, and will be correlated to irradiated fields. Calculated data for each study step will be compared in order to assess the extent of RT induced lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients both female and male above 18 years old referred to radiotherapy treatment of primary or secondary malignant involvement of the lung parenchyma.

Exclusion Criteria:

* Patients undergoing treatments that might induce lung toxicity other than the RT being assessed will be excluded.
* Patients suffering of lung illnesses as infection, pulmonary embolism, and congestive heart failure will be excluded.
* Special populations like pregnant women, children and legally incompetent patients will not be included in this study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-10 (Estimated); Primary Completion 2019-04-02 (Estimated); Study Completion 2020-04-02 (Estimated)

PRIMARY OUTCOMES:
Measuring the change of pulmonary function reserve in relation to the irradiated field, before and after treatment, using quantification software. | For the individual patient, the duration of participation is six months.
  The data will analysed using quantification software

IPD SHARING:
Plan to Share IPD: Undecided